CLINICAL TRIAL: NCT06188585
Title: Randomized Controlled Multi-Center Non-Inferiority Trial of UI-EWD (Nexpowder™) vs. Conventional Treatment as First-Line Endoscopic Therapy for Patients With High-Risk Nonvariceal Upper Gastrointestinal Bleeding (TREET)
Brief Title: Randomized Trial of UI-EWD vs. Conventional Endoscopic Therapy for Nonvariceal Upper Gastrointestinal Bleeding
Acronym: TREET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Collaborators: North American Science Associates Ltd. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDT23013
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-07

CONDITIONS: Acute Gastrointestinal Bleeding
Keywords: Gastrointestinal hemorrhage; Peptic Ulcer; Nonvariceal upper gastrointestinal bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Peptic Ulcer | interventions — Indicator Dilution Techniques; Injections; Argon Plasma Coagulation

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned with concealed allocation in a 1:1 ratio to receive treatment with UI-EWD hemostatic powder (Nexpowder) or conventional endoscopic hemostatic therapy (defined as bipolar electrocoagulation or clips or argon plasma coagulation with or without epinephrine injection therapy).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Test Group (Experimental): UI-EWD
  Interventions: Device: UI-EWD
- Control Group (Active Comparator): Conventional endoscopic therapy
  Interventions: Device: Conventional therapy

INTERVENTIONS:
Device: UI-EWD — Hemostatic powder administered at index endoscopy
  Other Names: Nexpowder™
  Arms: Test Group
Device: Conventional therapy — Conventional endoscopic therapy (bipolar electrocoagulation or clips or argon plasma coagulation, with or without epinephrine injection) administered at index endoscopy
  Other Names: Bipolar electrocoagulation or Bipolar electrocoagulation endoscopic hemostasis; Epinephrine (1:10,000 dilution) injection or Endoscopic hemostatic injection of epinephrine (1:10,000 dilution); Endoscopic hemostatic clip; Argon plasma coagulation
  Arms: Control Group

SUMMARY:
A prospective, multi-center, noninferiority randomized controlled trial designed to compare the efficacy of UI-EWD (Nexpowder™) hemostatic powder versus conventional endoscopic hemostatic therapy in patients presenting with acute overt gastrointestinal bleeding which is found at endoscopy to be due to one of the following sources: a gastric or duodenal ulcer with active bleeding (spurting or oozing) or a non-bleeding visible vessel; an esophageal, gastric or duodenal tumor with active bleeding or a non-bleeding visible vessel; a gastric or duodenal Dieulafoy lesion with active bleeding or a non-bleeding visible vessel; or an actively bleeding Mallory-Weiss tear.

DETAILED DESCRIPTION:
Endoscopic hemostatic therapy is recommended as the first line therapy for patients with upper gastrointestinal bleeding (UGIB) due to ulcers with active bleeding or a non-bleeding visible vessel identified at endoscopy. A variety of endoscopic modalities are used in the treatment of UGIB, including thermal therapies (e.g., bipolar electrocoagulation), injection therapy (e.g., epinephrine), clips, and hemostatic powder spray. Topical therapies, such as hemostatic powder spray, have been the most recent addition to the armamentarium of endoscopic therapies for UGIB.

UI-EWD hemostatic powder (Nexpowder™), which is manufactured by NextBiomedical and distributed by Medtronic, is approved for treatment of nonvariceal GI bleeding in the U.S., Canada, European Union and other countries.

A retrospective study of UI-EWD hemostatic powder in 56 patients with active bleeding found immediate hemostasis in 54 (96.4%), with rebleeding within 7 days in only 2 patients (3.7%)[1]. A large multi-center randomized trial in 340 patients with nonvariceal UGIB and either active bleeding or a non-bleeding visible vessel compared conventional endoscopic hemostatic therapy alone to conventional therapy plus UI-EWD. Rebleeding was significantly lower in the UI-EWD group at 3 days (3 vs. 11%) and at 30 days (19% vs. 7%) [2].

The primary aim of this trial is to demonstrate that UI-EWD when used as initial hemostatic therapy is non-inferior to older conventional endoscopic hemostatic therapy for the treatment of patients with high-risk nonvariceal upper GI bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 22 years or older
2. Presentation with acute overt gastrointestinal bleeding (hematemesis, melena, and/or hematochezia)
3. Subject voluntarily agrees to participate in the clinical investigation, provides written informed consent, and will be able to comply with the investigational protocol in the opinion of the site investigator
4. Cause of bleeding as determined at upper endoscopy is one of the following sources: a gastric or duodenal ulcer with active bleeding (spurting or oozing) or a non-bleeding visible vessel; an esophageal, gastric or duodenal tumor with active bleeding or a non-bleeding visible vessel; a gastric or duodenal Dieulafoy lesion with active bleeding or a non-bleeding visible vessel; or an actively bleeding Mallory-Weiss tear. The definition of "active oozing" will require bleeding to persist for ≥ 3 minutes of endoscopic observation.

Exclusion Criteria:

1. Incarceration
2. Subjects that are not able to provide written informed consent
3. Pregnancy or nursing mothers
4. Endoscopic hemostatic treatment in the past 30 days
5. Use of triple antithrombotic therapy at the time of presentation
6. Subjects who underwent gastric or duodenal endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) procedures within the past 2 months
7. Post-polypectomy bleeding
8. Subjects with erosive esophagitis, erosive gastritis, esophageal ulcer, or vascular ectasia including gastric antral vascular ectasia
9. Platelet count < 50 x 10^9/L
10. INR > 3.5 (or prothrombin time >35 seconds in patient not on warfarin and only prothrombin time is provided by local lab), at time of procedure or closest to procedure time
11. Subjects who have documented galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
12. Subjects with documented hypersensitivity to Brilliant Blue FCF
13. Subjects with suspected bowel obstruction or gastrointestinal fistulas, and those suspected or are at high risk of having gastrointestinal perforation.
14. Endoscopy not performed within 36 hours of presentation to hospital/emergency department

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
No further bleeding during the 7-day period after hemostatic treatment | 7 days
  Further bleeding includes patients with persistent bleeding despite study-assigned endoscopic therapy or patients with recurrent bleeding

SECONDARY OUTCOMES:
Composite 30-day outcome of further bleeding | 30 days
  Further bleeding leading to red blood cell transfusion or urgent intervention (need for alternative therapy at index endoscopy, repeat endoscopy, interventional radiology, or surgery)
Initial hemostasis for patients with active bleeding at randomization | During index endoscopy procedure
  Initial hemostasis with study-assigned endoscopic therapy for patients with active bleeding
Number of participants with recurrent bleeding over the 7-day period after randomization | 7 days
  Recurrent bleeding among all patients with hemostasis within 7 days after study-assigned endoscopic therapy
Mortality | 30 days
  30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Loren Laine, MD, Study Chair — Yale University
Locations (15):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - Yale, New Haven, Connecticut
  - RUSH University, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Rutgers University, Piscataway, New Jersey
  - Northwell Health, Manhasset, New York
  - NYU Langone, New York, New York
- Canada (3):
  - McGill University, Montreal, Quebec
  - St. Michael's Hospital, Toronto
  - Vancouver General Hospital, Vancouver
- Denmark (2):
  - Copenhagen University Hospital, Hvidovre
  - Odense University Hospital, Odense
- St. Antoine, Paris, France
- Emek Medical Center, Afula, Israel
- Cleveland Clinic London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park JS, Kim HK, Shin YW, Kwon KS, Lee DH. Novel hemostatic adhesive powder for nonvariceal upper gastrointestinal bleeding. Endosc Int Open. 2019 Dec;7(12):E1763-E1767. doi: 10.1055/a-0982-3194. Epub 2019 Dec 10. PMID 31828214
- [Background] Cha B. A Randomized Control Study Evaluating the Efficacy of a Hemostatic Powder (UI-EWD) in Decreasing the Rate of Upper Gastrointestinal Re-Bleeding in Patients Treated with Endoscopic Therapy for High-Risk Lesions. Oral presentation presented at: Digestive Disease Week 2023; May 9, 2023; Chicago, IL.
- [Derived] Al Alawi S, Bessissow T, Fallone CA, Jacques J, Barkun A. Hemostatic powder's battle against a spurting bleeding ulcer: can it win? Endoscopy. 2025 Dec;57(S 01):E676-E677. doi: 10.1055/a-2610-3096. Epub 2025 Jun 26. No abstract available. PMID 40570926